CLINICAL TRIAL: NCT01635309
Title: Coronary CT Angiography to Predict Vascular Events In Noncardiac Surgery patIents cOhort evaluatioN (CTA -VISION) Study
Acronym: CTA-VISION
Status: Completed | Type: Observational
Sponsor: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Philip Devereaux, Principal Investigator, McMaster University
Organization: McMaster University (Other)
Other Study IDs: CTA-VISION
Record Dates: First submitted 2012-07-04; First posted 2012-07-09 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Non-cardiac surgical patients: >= 45 years old, undergoing non-cardiac surgery requiring regional or general anaesthetic and an overnight stay with cardiac risk factors
  Interventions: Other: Coronary CT Angiogram

INTERVENTIONS:
Other: Coronary CT Angiogram — pre-operative coronary CTA

SUMMARY:
Worldwide 200 million adults annually undergo major noncardiac surgery and 5 million of these patients will suffer a major vascular complication. Despite the magnitude of this problem our capacity to predict these events is limited. Although perioperative myocardial infarction (MI) is the most common major perioperative cardiac complication, little is known about its pathophysiology. Coronary computed tomography angiography (CTA) is a potential non-invasive method for the detection of coronary artery disease and cardiac risk stratification in the non-operative setting; however, the value of this test to enhance risk prediction among patients scheduled for noncardiac surgery is unknown. This study is an international prospective cohort study to determine among patients with, or at risk of, atherosclerotic disease who are undergoing noncardiac surgery: 1) if preoperative coronary CTA has additional predictive value for the occurrence of major perioperative cardiac events and 2) the underlying coronary anatomy associated with perioperative MIs.

ELIGIBILITY:
Inclusion Criteria:

* age >=45 years
* undergoing non cardiac surgery requiring an overnight stay and general or regional anaesthetic
* at least one of:

  1. Coronary Artery Disease (CAD)
  2. Peripheral Vascular Disease (PVD)
  3. History of Stroke
  4. History of Congestive Heart Failure (CHF)
  5. Combination of at least 3 of:
* age >= 70 years
* history of treatment for hypertension
* history of treatment for dyslipidemia
* smoking in last 2 years
* diabetic and currently taking insulin or oral diabetic drugs
* history of Transient Ischemic Attack (TIA)

Exclusion Criteria:

* contraindications to CTA

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: International non cardiac surgical patients
Sampling Method: Non-Probability Sample
Enrollment: 987 (Actual)
Dates: Start 2007-05; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Perioperative MI | 30-days post-operative

SECONDARY OUTCOMES:
Perioperative Cardiovascular Event | 30-days post-operative

CONTACTS AND LOCATIONS:
Locations (1):
- Juravinski Hospital, Hamilton, Ontario, Canada

REFERENCES:
- [Result] Sheth T, Chan M, Butler C, Chow B, Tandon V, Nagele P, Mitha A, Mrkobrada M, Szczeklik W, Faridah Y, Biccard B, Stewart LK, Heels-Ansdell D, Devereaux PJ; Coronary Computed Tomographic Angiography and Vascular Events in Noncardiac Surgery Patients Cohort Evaluation Study Investigators. Prognostic capabilities of coronary computed tomographic angiography before non-cardiac surgery: prospective cohort study. BMJ. 2015 Apr 22;350:h1907. doi: 10.1136/bmj.h1907. PMID 25902738
- [Derived] Walpot J, Massalha S, Jayasinghe P, Sadaf M, Clarkin O, Godkin L, Sharma A, Ratnayake I, Godkin K, Jia K, Hossain A, Crean AM, Chan M, Butler C, Tandon V, Nagele P, Woodard PK, Mrkobrada M, Szczeklik W, Aziz YFA, Biccard B, Devereaux PJ, Sheth T, Chow BJW. Normalized Subendocardial Myocardial Attenuation on Coronary Computed Tomography Angiography Predicts Postoperative Adverse Cardiovascular Events: Coronary CTA VISION Substudy. Circ Cardiovasc Imaging. 2022 Jan;15(1):e012654. doi: 10.1161/CIRCIMAGING.121.012654. Epub 2022 Jan 18. PMID 35041449